CLINICAL TRIAL: NCT00087074
Title: A Trial of CCI-779 in Patients With Soft Tissue Sarcoma.
Brief Title: CCI-779 in Treating Patients With Soft Tissue Sarcoma or Gastrointestinal Stromal Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02809; MC027B; N01CM17104 (NIH)
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Gastrointestinal Stromal Tumor; Recurrent Adult Soft Tissue Sarcoma; Stage I Adult Soft Tissue Sarcoma; Stage II Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Sarcoma | interventions — temsirolimus; Sirolimus

ARMS (1):
- Treatment (temsirolimus) (Experimental): Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 additional courses beyond CR.
  Interventions: Drug: temsirolimus; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase II trial is studying how well CCI-779 works in treating patients with soft tissue sarcoma or gastrointestinal stromal tumor. Drugs used in chemotherapy, such as CCI-779, work in different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the antitumor activity of CCI-779 in this patient population.

SECONDARY OBJECTIVES:

I. To assess the following in patients with soft tissue sarcomas and following treatment with CCI-779: duration of response, time to progression, survival.

TERTIARY OBJECTIVES:

I. To describe and correlate the following with patient characteristics and outcome in this patient population and following treatment with CCI-779: relative levels of 4EBP1 to eIF4E, phospho 4EBP1, total and phospho ribosomal S6 on pretreatment tumor tissue, expression levels of EGFR, activated EGFR, Her2, c-Myc, phospho Akt, total Akt, phospho-mTOR and total mTOR on pretreatment tumor tissue, drug induced inhibition of p70S6 kinase activity, and phosphorylation of S6 in PBMC, relative levels of serum sirolimus in post-treatment samples.

OUTLINE:

Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 additional courses beyond CR.

Patients are followed every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologic confirmed soft tissue sarcoma
* Measurable disease; for patients having only lesions measuring at least 1 cm to less than 2 cm, must use spiral CT imaging for both pre- and post-treatment tumor assessments
* Absolute neutrophil count (ANC) >= 1,500/μL
* Platelets (PLTS) >= 100,000/μL
* Hgb >= 10.0 g/dL
* Direct bilirubin =< 1.5 x ULN (upper limit normal)
* AST(SGOT) =< 2.5 x ULN or =< 5 x ULN* if liver metastases are present
* ALT(SGPT) =< 2.5 x ULN or =< 5 x ULN* if liver metastases are present
* Creatinine =< 1.5 x ULN, or if greater, creatinine clearance >= 50 mL/min/1.73 m^2
* Baseline glucose levels
* Fasting serum cholesterol =< 350 mg/dL (9.0 mmol/L)
* Fasting triglycerides =< 400 mg/dL (4.56 mmol/L)
* ECOG Performance Status (PS) 0, 1 or 2
* Life expectancy >= 12 weeks
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent

Exclusion Criteria:

* Any of the following as this regimen may be harmful to a developing fetus or nursing child:

  * Pregnant women
  * Breast-feeding women
  * Men or women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception ( diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.)
* Any of the following:

  * Nitrosoureas or mitomycin =< 6 weeks prior to study entry
  * Other chemotherapy =< 4 weeks prior to study entry
  * Radiotherapy =< 4 weeks prior to study entry
  * Concurrent use of any other investigation agent
  * Adverse events due to agents administered =< 4 weeks prior to study entry
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CCI-779
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, diabetes, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known HIV-positive patients receiving combination anti-retroviral therapy
* Prior chemotherapy for metastatic disease

  * Exceptions:

    * Patients with GIST who fail Gleevec are eligible
    * Patients who have had adjuvant/neoadjuvant chemotherapy are also eligible
* Known brain metastases

  * Exception: Patients with treated brain metastatic disease with stable symptoms after treatment for >= 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2004-06; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Proportion of confirmed tumor responses, defined to be either a CR or PR noted as the objective status on 2 consecutive evaluations at least 4 weeks apart | Up to 6 months (6 courses)

SECONDARY OUTCOMES:
Survival time | Time from registration to death due to any cause, assessed up to 5 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time to disease progression | Time from registration to documentation of disease progression, assessed up to 5 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Duration of response is defined for all evaluable patients who have achieved an objective response as the date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented | Up to 5 years
Time to treatment failure | Time from the date of randomization to the date at which the patient is removed from treatment due to progression, toxicity, or refusal, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott Okuno, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States